CLINICAL TRIAL: NCT06113679
Title: EB-PCC-01, A Pilot Randomized, Sham Controlled Safety and Efficacy Study of the EmitBio™ RD-X19 Treatment Device in Subjects With Post COVID-19 Condition (PCC) in the Outpatient Setting
Brief Title: Pilot Randomized Study of RD-X19 Tx Device in Subjects With PCC (Long Covid) in the Outpatient Setting
Acronym: EB-PCC-01
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment stopped by Sponsor following interim analysis data review.
Sponsor: EmitBio Inc. (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Organization: KNOWBio Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EB-PCC-01; Pro00074175 (Other: Advarra IRB)
Record Dates: First submitted 2023-10-30; First posted 2023-11-02 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Post COVID-19 Condition (PCC)

STUDY DESIGN:
Intervention Model Description: Randomized, 1:1 Sham Control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Active (Active Comparator)
  Interventions: Device: RDX-19
- Sham (Sham Comparator)
  Interventions: Device: RDX-19

INTERVENTIONS:
Device: RDX-19 — RD-X19 device with a 5 minute, 32 J/cm2 dose, 2X/day, 7 days. Each treatment at least 6 hours apart.

SUMMARY:
Duration of Treatment: 7 days, 2 times per day.

Following Randomization on Week 1 Day 1, Subjects will continue to have televisits and rate symptoms and upright activity weekly during a 5 week follow up. Subjects will be followed via in clinic visits at week 2/day 8 (+3/-0 days) and Week 6 / day 36, (+3/-3days). Subjects will receive a weekly televisit during Week 3 / day 15 (+3/-3), Week 4 / day 22 (+3/-3), and Week 5 / day 29 (+3/-3).

DETAILED DESCRIPTION:
Subjects who have been pre-screened will be approached regarding the study and scheduled for a Screening Visit (V0). During the Screening Visit (V0) subjects will be consented and screened. To be considered eligible, subjects must present evidence of prior SARS-CoV-2 infection or COVID-19 via in clinic testing. Subject screening will include symptom assessments, medical history, and collection of laboratory samples. Following receipt of subject lab results, subjects who meet inclusion/exclusion criteria will be scheduled for Visit 1. At V1 eligible subjects will be randomized 1:1 to receive device or sham. Randomization will be performed.

During V1 which is Day 1 of treatment, subjects will receive in clinic training on the use of the device. Subjects will administer the first treatment while supervised in the clinic. The second treatment on Day 1 will be at home via a televisit performed by eligible clinical site staff.

At V1 subjects will identify and grade symptoms on a 4 point scale for both primary and secondary PCC symptoms. This evaluation will serve as a baseline for subsequent comparative assessments using the Patients Global Impression of Change 1(PGIC-1) scale.

After the first in clinic treatment, subjects will self treat at home during a prescheduled televisit. Televisits may be performed via web based telehealth applications or telephone with eligible clinical site staff. At each televisit, subjects will be asked questions regarding possible side effects and adverse events. Daily during the telehealth visit that occurs during treatment, clinical site staff will assess symptoms using the PGIC 1 scale and will assess their hours of upright activity..

Follow up will be performed for 5 weeks after treatment completion. During follow up telehealth visits subjects will be asked about any symptomswhich will include the PGIC 1 assessment and hours of upright activity.

At follow up week 2 (day 8 +3/- 0 days) subjects will return to the clinic for in person visual and physical health assessments, changes since last visit, safety assessments, and a blood draw. During the in clinic visit the subject will complete the PGIC 1 assessment and hours of upright activity assessment.

During weeks 3, 4, and 5, subjects will be followed via televisits, with each visits cheduled on approximately the same day each week. During the televisits, subjects will be asked questions regarding adverse events, the PGIC-1 assessment and hours of upright activity assessment will be performed..

At follow up week 6 (+/-3 days), subjects will return to the clinic for in person visual and physical health assessments, changes since last visit, safety assessments, and a blood draw. While in clinic, subjects will complete the final PGIC 1 scale, the PGIC 2 scale, and upright activity assessments. The PGIC 2 assessment is additional data not associated with an endpoint. Subjects will return the study devices..

Additional data collected as a part of the study will be the measure of cytokines and chemokines before and after treatment. Hours of upright activity over the course of the study will also be reported.. Both of these assessments are reported measures but are not associated with objectives or endpoints.

ELIGIBILITY:
Inclusion Criteria:

A subject must meet all the following criteria to be eligible for inclusion in this study:

1. History of confirmed diagnosis of SARS-CoV-2 infection or COVID-19 per section 9.4.
2. PCC (per protocol definition) with cough and at least 2 of the 3 additional qualifying symptoms that have been determined not associated with another disease state:

   * fatigue
   * shortness of breath
   * cognitive dysfunction/brain fog.
3. Negative for COVID-19 via rapid antigen test.
4. Minimum time period from onset of symptoms (or from date of positive test for asymptomatic) - 3 months.
5. Minimum duration of symptoms at least 2 months, continuous or intermittent.
6. Males or females, 22 years of age and older on the date of enrollment.
7. Provides written informed consent prior to initiation of any study procedures.
8. Be able to understand and agrees to fully comply with defined and described study procedures and be available for all study visits for the entire study duration.
9. Agrees to perform self-treatment twice a day, separated by ≥ 6 hours during the treatment period.
10. Agrees to maintain current medications without the addition of any new medications for relief of signs and symptoms of PCC during the entire study period, and, if used, to report ALL such medications (including over the counter and home remedies) to the study staff.
11. No uncontrolled disease process (chronic or acute) that could be attributable to qualifying symptoms.
12. No physical or mental conditions or attributes at the time of screening, which in the opinion of the PI, will prevent full adherence to, and completion of, the protocol.
13. For women of childbearing potential, a negative urine pregnancy test at screening. Subjects (female subjects of childbearing potential and male subjects with partners of childbearing potential) must agree to use proper** contraceptive methods to avoid pregnancy during the study.

Exclusion Criteria:

A subject with any of the following criteria will be excluded from participation in this study:

1. Positive test for SARS-CoV-2 infection or COVID-19 within the past 30 days.
2. Individuals < age 22 at consent.
3. Any medical disease or condition that, in the opinion of the site Principal Investigator (PI) or appropriate sub-investigator, precludes study participation.
4. History of recurrent alcohol intoxication or other recreational drug use (excluding medically prescribed cannabis) within 30 days of study day, V1.
5. History of any systemic antiviral therapies within 30 days of study day, V1.
6. History of oral or parenteral corticosteroid use within 30 days of study day, V1. Active use of nasal or inhalable corticosteroids is also exclusionary. Topical steroids are not exclusionary.
7. History of any chronic medical condition that has required adjustments to the type, dose, or schedule of medical treatments within 30 days of study day, V1.
8. Requirement to use narcotic medication for analgesia.
9. History of hypersensitivity or severe allergic reaction (e.g., anaphylaxis, generalized urticaria, angioedema, other significant reaction) to sun exposure.
10. Presence of any oral abnormality (e.g., including, but not limited to, ulcer, oral candidiasis, oral mucositis, gingivitis, history of frequent recurrent aphthous ulcers, burning mouth syndrome, dry mouth syndrome, a disease that can result in xerostomia (e.g., Sjogren's syndrome), or other oral disorder that in the opinion of the investigator would interfere with device use and evaluation.
11. Any intra-oral metal body piercings that cannot be removed for the duration of the study. Metal orthodontia is permitted as braces will be covered by the device mouthpiece.
12. Any individual without teeth or with a dental malformation that precludes directed use of the device as intended.
13. Use of new medications to treat PCC symptoms within the 30 days prior to V1.
14. Currently enrolled in or plans to participate in another clinical trial with a therapeutic investigational agent for any medical indication that will be received during the study period.
15. Has participated in an investigational treatment trial for PCC within the past 30 days.
16. Subjects with immunodeficiency syndromes, including HIV, per medical history diagnosed prior to previous acute COVID-19.
17. Subjects who have previously participated in RD-X19 acute studies, P20 or P30.
18. Is pregnant or nursing, is not post-menopausal, or is not currently on birth control. The rhythm method is not an acceptable form of birth control for this study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Primary Symptom Improvement | 5 weeks
  Improvement of one or more primary PCC signs/symptom(s) - cough, fatigue, shortness of breath, cognitive dysfunction/brain fog as compared to sham, with or without fluctuation.

SECONDARY OUTCOMES:
Secondary Symptom Improvement | 5 weeks
  Improvement of one or more secondary PCC signs/symptoms as compared to sham, with or without fluctuation:
  * chest pain
  * altered smell/taste
  * headache
  * joint pain
  * muscle pain/spasms
  * post exertional malaise
  * sleep disorders
  * tachycardia/palpitations,and
  * GI/abdominal symptoms (include but not limited to abdominal pain, nausea, diarrhea, vomiting).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Site 2_WellNow Urgent Care and Research, East Amherst, New York
  - Site 1_Helios - Physician Quality Care, Milan, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided